CLINICAL TRIAL: NCT01618331
Title: The Effect of Protein Supplementation Doing Regular Exercise in Patients With Facioscapulohumeral Muscular Dystrophy - a Blinded RCT Study
Brief Title: Protein Supplementation and Exercise in Patients With FSH Muscular Dystrophy- a Randomized Placebo Controlled Study
Acronym: FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grete Andersen, MD (Other)
Collaborators: The Augustinus Foundation, Denmark. (Other); Aase and Ejnar Danielsens Foundation (Other); The Danish Rheumatism Association (Other); AP Moeller Foundation (Other)
Responsible Party: Sponsor-Investigator, Grete Andersen, MD, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-1-2011-149
Record Dates: First submitted 2012-06-07; First posted 2012-06-13 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Facioscapulohumeral Muscle Dystrophy
Keywords: FSHD; Endurance exercise; Protein supplementation; Placebo RCT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein supplementation (Active Comparator): Patients consume a drink after each exercise session. The drink consist of whey protein, maltodextrin, and flavors mixed in water.
  Interventions: Behavioral: Regular exercise; Dietary Supplement: Protein-carbohydrate supplementation
- Placebo supplement (Placebo Comparator): Patients consume a drink after each exercise session. The drink consist of flavors mixed in water.
  Interventions: Behavioral: Regular exercise
- Control (No Intervention): Patients will be tested before and after a none-intervention period of 12 weeks.

INTERVENTIONS:
Behavioral: Regular exercise — Duration: 3 session each week, in 12 week. Intensity: 70 % of VO2max. Type: cycle-ergometer exercise.
  Arms: Placebo supplement; Protein supplementation
Dietary Supplement: Protein-carbohydrate supplementation — Dosage: 45g powder mixed in 0.5 L water After each exercise session, 3 times each week, in 12 weeks.
  Arms: Protein supplementation

SUMMARY:
The hypotheses is that regular post exercise supplementation increase fitness and daily activity level in patients with Fascioscapulohumeral (FSH) muscular dystrophy.

All patients are tested before and after 12 weeks of cycle-ergometer exercise. Maximal oxygen consumption and 6MWT is used as primarily effect goals. Secondary effect goals are risk of falls and daily activity level.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the response to protein-carbohydrate supplementation doing regular exercise in patients with FSHD. All patients are tested before and after 12 weeks of cycle-ergometer exercise. Maximal oxygen consumption and a functional 6 min walk test(6MWT) is used as primarily effect goals. Secondary effect goals are risk of falls and daily activity level. We measure manuel muscle strength, a balance test, a 5-time-up-and-down-chair-test, a 14 steps-stair-test, accelerometer measuring, daily activity level questionnaire and SP36.

We use a blinded randomized controlled trail. The interventions are 12 weeks regular exercise and consumption of a post-exercise drink. The exercise consists of 30 session of 30 minutes moderate exercise on a cycle-ergometer. After each exercise session patients consume a protein or a non-caloric placebo drink.

ELIGIBILITY:
Inclusion Criteria:

* Verified FSHD
* Age 18-65
* Untrained. Less than two hours cardio-training each week the last 4 month.

Exclusion Criteria:

* Competitive disorders
* Pregnant and breastfeeding
* Unable to walk 200 m within 6 min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption test | up to Week 12
  All participant are tested with a standardized maximal oxygen consumption test. Maximal oxygen uptake pr. minute pr. kg body (VO2max) weight and maximal work load (Wmax) is measured. The effect of intervention is found in different between groups in relative and absolute improvement in VO2max and Wmax.
6MWT | up to Week 12
  6 min walk test. Outcome in meter.

SECONDARY OUTCOMES:
Risk of falls | week: 0 and 12
  Measuring of: Muscle strength, balance, 5-times-up-and-down-chair-test, 14-steps-stair-test.
Daily activity level | week: 0 and 12
  assessment of daily-activity level by accelerometer daily-activity level questionary SP36 life quality questionary
Blood samples | week: 0, 4, 7, 10, 12
  Creatine Kinase and myoglobin levels (safe parameter) Inflammatory level

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, Department of Neurology, Rigshospitalet, Copenhagen, Denmark